CLINICAL TRIAL: NCT05737849
Title: To Investigate EGFR Exon20 Insertion Mutation Testing Methodologies, Clinicopathological Characteristics and Molecular Epidemiology in Chinese Patients With Advanced NSCLC: a Nationwide Multicentre Real-world Registry Study
Brief Title: A Study to Learn About the Tests Looking for a Gene Mutation in Adults With Lung Cancer in China (ELEGANT)
Acronym: ELEGANT
Status: Withdrawn | Type: Observational
Why Stopped: Business reason, unrelated to product safety
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-788-4004
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: Drug Therapy; EGFR exon20 insertion mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Participants With Positive EGFR ex20ins Detection: Participants with NSCLC having positive EGFR ex20ins detected by NGS were observed retrospectively for three years prior to leading site initiation.
  Interventions: Other: No Intervention
- Cohort 2: Participants With Positive and Negative EGFR ex20ins Detection: Participants with NSCLC having positive and negative EGFR ex20ins NGS testing results were observed retrospectively for three years prior to leading site initiation.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — As this is an observational study, no intervention will be administered in this study.

SUMMARY:
The main aim of this study is to examine the percentage of people with lung cancer who carry a certain gene mutation (epidermal growth factor receptor exon 20 insertions - EGFR ex20ins) and their frequency in Chinese participants with Non-small cell lung cancer (NSCLC) after having been tested for the gene mutation.

Data from the participant's electronic medical records at the hospital will be collected.

DETAILED DESCRIPTION:
This is a non-interventional, retrospective, observational study of the Chinese participants with locally advanced or metastatic NSCLC with EGFR ex20ins mutation. The primary objective of this study is to explore the prevalence of EGFR ex20ins, subtypes of EGFR ex20ins and their frequency in Chinese participants with locally advanced or metastatic NSCLC.

The study will enroll approximately 10800 patients. Participants will be enrolled in the following two cohorts:

* Cohort 1: Participants With Positive EGFR ex20ins Detection
* Cohort 2: Participants With Positive and Negative EGFR ex20ins Detection

The data will be collected retrospectively using the participant electronic medical records and next-generation gene sequencing (NGS)/polymerase chain reaction (PCR) kit instructions.

This multi-center trial will be conducted at 15 sites across China. The overall time to participate and data collection will be approximately 12 months.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1 and 2:

1. Participants with a diagnosis of locally advanced or metastatic NSCLC, clinical staging of IIIB-IV.

Cohort-1:

1. Participants who have received NGS testing and have EGFR ex20ins positive result.

Cohort-2:

1. Participants who have received NGS testing

Exclusion Criteria:

1. Incomplete information, including key demographic characteristics, clinicopathological characteristics, and genetic testing information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort 1: Participants with locally advanced or metastatic NSCLC who received NGS testing and have EGFR ex20ins positive results.
  Cohort 2: Participants with locally advanced or metastatic NSCLC who received NGS testing.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-01-30 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Cohort 2: Prevalence of EGFR ex20ins in Chinese Participants With Locally Advanced or Metastatic NSCLC | Up to 3 years prior to leading site initiation
  The prevalence of EGFR ex20ins will be reported for participants with locally advanced or metastatic NSCLC.
Cohort 1 and 2: Number of EGFR ex20ins Subtypes in Chinese Participants With Locally Advanced or Metastatic NSCLC | Up to 3 years prior to leading site initiation
  EGFR ex20ins subtype is defined by insertion or duplication mutation occurred in amino acids (AA) 761 to AA775 of EGFR gene. The number of EGFR ex20ins subtypes will be reported.
Cohort 1 and 2: Frequency of Each EGFR ex20ins Subtype in Chinese Participants With Locally Advanced or Metastatic NSCLC | Up to 3 years prior to leading site initiation
  The frequency of each EGFR ex20ins subtype will be reported.

SECONDARY OUTCOMES:
Cohort 1 and 2: Percentage of Theoretically Underdiagnosed EGFR ex20ins Mutation by Different PCR Kits Based on NGS Real-world Database | Up to 3 years prior to leading site initiation
  The theoretically underdiagnosed rate about EGFR ex20ins detection by different PCR kits available in China will be reported.
Cohort 1 and 2: Number of EGFR ex20ins Positive Participants With Demographic Characteristics | Up to 3 years prior to leading site initiation
  Demographic characteristics include age, gender, smoking history and family history for malignancies.
Cohort 1 and 2: Number of EGFR ex20ins Positive Participants With Clinical Stages of Lung Cancer at the Time of NGS Testing | Up to 3 years prior to leading site initiation
  Number of EGFR ex20ins positive participants with the clinical stages of cancer IIIB, IIIC, IV will be evaluated using the international association for the study of lung cancer eighth edition of the tumor, nodes, and metastases (TNM) classification for staging criteria.
Cohort 1 and 2: Number of EGFR ex20ins Positive Participants With Cytology or Histology at the Time of NGS Testing | Up to 3 years prior to leading site initiation
  Number of EGFR ex20ins positive participants with adenocarcinoma, squamous cell carcinoma, mixed, or other carcinomas will be evaluated.
Cohort 1 and 2: Site of Metastasis at the Time of NGS Testing | Up to 3 years prior to leading site initiation
  Site of metastasis at the time of NGS testing will be reported.
Cohort 1 and 2: Number and Kinds of Co-occurring Mutations of EGFR ex20ins at Baseline in Positive Participants Detected by NGS Testing | Baseline (prior to NGS testing)
  The number and kinds of co-occurring mutations at baseline will be reported. The baseline is defined as treatment naive before NGS testing.
Cohort 2: Number of EGFR ex20ins Positive Participants, Participants With Common EGFR Mutations and Participants With EGFR Wild Type With Demographic Characteristics | Up to 3 years prior to leading site initiation
  Demographic characteristics include age, gender, smoking history and family history for malignancies.
Cohort 2: Number of EGFR ex20ins Positive Participants, Participants With Common EGFR Mutations and Participants With EGFR Wild Type With Clinical Stages of Lung Cancer at the Time of NGS Testing | Up to 3 years prior to leading site initiation
  Number of EGFR ex20ins positive participants, participants with common EGFR mutations and participants with EGFR wild type with the clinical stages of cancer IIIB, IIIC, IV will be evaluated using the international association for the study of lung cancer eighth edition of the TNM classification for staging criteria.
Cohort 2: Number of EGFR ex20ins Positive Participants, Participants With Common EGFR Mutations and Participants With EGFR Wild Type With Cytology or Histology at the Time of NGS Testing | Up to 3 years prior to leading site initiation
  Number of EGFR ex20ins positive participants, participants with common EGFR mutations and participants with EGFR wild type with adenocarcinoma, squamous cell carcinoma, mixed, or other carcinomas will be evaluated.
Cohort 2: Site of Metastasis at the Time of NGS Testing | Up to 3 years prior to leading site initiation
  Site of metastasis at the time of NGS testing will be reported.
Cohort 2: Number and Kinds of Co-occurring Mutations at Baseline in EGFR ex20ins Positive Participants, Participants With Common EGFR Mutations and Participants With EGFR Wild Type Detected by NGS Testing | Baseline (prior to NGS testing)
  The number and kinds of co-occurring mutations at baseline will be reported. The baseline is defined as treatment naive before NGS testing.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Department of Pathology, National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences (CAMS) and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/1d4babd8980d494d?idFilter=%5B%22TAK-788-4004%22%5D